CLINICAL TRIAL: NCT05756608
Title: Fibrosis in Chronic and Delayed Myocardial Infarction
Acronym: FCDMI
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 300754
Record Dates: First submitted 2023-02-18; First posted 2023-03-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Aortic Stenosis; Chemotherapy Induced Systolic Dysfunction; Carcinoid Syndrome
MeSH Terms: conditions — Aortic Valve Stenosis; Serotonin Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aortic stenosis: The investigators will recruit 70 patients with aortic stenosis (25 patients with asymptomatic moderate aortic stenosis and 25 patients with symptomatic severe aortic stenosis, 10 patients with mild aortic stenosis and 10 patients with aortic sclerosis) and 10 healthy volunteers, who will undergo baseline 68Ga-FAPI or 18F-AlF-FAPI PET/MR imaging to establish fibrosis activity in healthy myocardium and in context of chronic myocardial injury. All patients will have a follow up FAPI PET/ MR scan 1 year after their baseline scan to assess whether myocardial fibrosis activity reverses following aortic valve replacement and restoration of normal afterload in patients with severe aortic stenosis and if baseline myocardial fibrosis activity can predict progression in the fibrosis burden and clinical progression in patients with mild or moderate aortic stenosis or aortic sclerosis. Healthy volunteers will not undergo any repeat imaging.
  Interventions: Diagnostic Test: 68Ga-FAPI and 18F-AlF-FAPI PET-MR
- Chemotherapy-induced cardiotoxicity: The investigators will recruit 60 patients who have undergone anthracycline treatment >1 year from enrollment and 10 healthy volunteers as part of this cohort. This will include 50 patients who have either clear evidence of cardiotoxicity (Ejection fraction <50% and a 10%point fall in ejection fraction) or a subclinical cardiac injury (elevated troponin, elevated T2, impaired global longitudinal strain) and 10 patients with no evidence of cardiotoxicity on their cardiac MRI scan (performed as part of the ongoing Cardiac CARE study). These patients will undergo baseline FAPI PET/MR imaging to establish the extent and pattern of myocardial fibrosis activity in context of delayed myocardial injury (chemotherapy-induced cardiotoxicity). All patients will have a follow up cardiac MRI scan 1-2 years after their baseline scan to assess whether baseline fibrosis activity is associated with a deterioration in cardiac function. Healthy volunteers will not undergo any repeat imaging.
  Interventions: Diagnostic Test: 68Ga-FAPI and 18F-AlF-FAPI PET-MR
- Carcinoid syndrome: In collaboration with the South East Scotland NET Service, the investigators will recruit 30 patients with carcinoid syndrome for this cohort. These patients will undergo a baseline echocardiogram and a FAPI PET/MR scan to investigate fibrosis activity within the cardiac chambers and valves. The investigators will recruit patients with established cardiac involvement as well as carcinoid syndrome patients with high circulating 5-HT concentrations who have no evidence of valve disease on echocardiography. All patients will have a follow up cardiac MRI scan and an echocardiogram, 6 months - 1 year after their baseline scan to assess whether baseline fibrosis activity is associated with subsequent deterioration in cardiac and valvular function.
  Interventions: Diagnostic Test: 68Ga-FAPI and 18F-AlF-FAPI PET-MR

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI and 18F-AlF-FAPI PET-MR — Hybrid Cardiac PET-MR with 68Ga-FAPI and 18F-AlF-FAPI radiotracer

SUMMARY:
In this study the investigators aim to examine the role that fibrosis plays in heart conditions such as aortic stenosis , chemotherapy-induced cardiotoxicity and carcinoid syndrome . Fibrosis is a common final result following any injury to the heart muscle and the investigators aim to identify this process early and in its active state. This will be examined by using a radiotracer 68Ga-FAPI or 18F-AlF-FAPI and PET-MRI or PET-CT.

DETAILED DESCRIPTION:
The investigators aim to investigate the role of fibrosis activity using 68Ga-FAPI and 18F-AlF-FAPI PET in chronic and delayed valvular, myocardial and endocardial injury states, in particular aortic stenosis, chemotherapy induced cardiotoxicity and carcinoid heart disease. The investigators also aim to analyse serum markers of myocardial injury and fibrosis at different time-points in these patient cohorts.

Research Hypothesis

1. In patients with aortic stenosis, myocardial fibrosis activity will correlate with markers of left ventricular decompensation and aortic valve fibrosis activity, will predict progression in fibrosis burden and will decline following aortic valve replacement.
2. Increased myocardial fibrosis activity will be observed in the early stages of anthracycline- induced cardiotoxicity and will predict later deterioration in cardiac function.
3. In patients with carcinoid syndrome, increased endocardial fibrosis activity will be observed in patients with subclinical and clinically significant valve involvement.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1(Aortic stenosis):

* Male or female above the age of 50 years old
* Provision of informed consent prior to any study specific procedures
* 25 patients with symptomatic severe aortic stenosis (peak velocity >4.0 m/s)
* 25 patients with moderate aortic stenosis (peak velocity 3.0-4.0 m/s)
* 10 patients with mild aortic stenosis (peak velocity 2.6-2.9 m/s)
* 10 patients with aortic sclerosis (tri-leaflet thickened aortic valve with no obstruction of ventricular outflow)
* 10 healthy volunteers (no other significant co-morbidities, as assessed by the study PI)

Cohort 2 (Chemotherapy-induced cardiotoxicity):

* Male or female over the age of 35 years with evidence of cardiotoxicity on cardiac MRI (performed as part of the Cardiac care study), at least 1 year after anthracycline treatment.
* 10 patients over the age of 35 years (male or females) without evidence of fibrosis on their 1-year scan after anthracycline treatment.
* 10 healthy volunteers (>35 years of age) with no significant co-morbidities, as assessed by the study PI.
* Provision of informed consent prior to any study specific procedures

Cohort 3 (Carcinoid syndrome):

* 30 patients with carcinoid syndrome (with or without cardiac involvement), over the age of 35 years, diagnosed as per consensus guidelines
* Provision of informed consent prior to any study specific procedures

Exclusion Criteria:

* Inability or unwilling to give informed consent.
* History of claustrophobia or feeling of inability to tolerate supine position for the MRI scans.
* Impaired renal function with eGFR of <30 mL/min/1.73m2.
* Women who are pregnant or breastfeeding.
* Contrast allergy
* Contraindication to cardiac MRI (e.g. metallic implant or severe claustrophobia)
* Recent myocardial infarction, other known causes of cardiomyopathy/cardiac fibrosis.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1: 70 patients with aortic stenosis with 10 matched healthy volunteers Cohort 2: 60 patients with Chemotherapy-induced cardiotoxicity and 10 healthy volunteers Cohort 3: 30 patients with carcinoid syndrome
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Fibrosis activity: Standardised uptake values (SUV | 1-2 years
  SUV
Fibrosis activity:Tissue-to-Background Ratio | 1-2 years
  TBR

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dweck, MBBS PhD, Study Chair — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided